CLINICAL TRIAL: NCT02850783
Title: Sentinel Lymph Node Identification in Colon Cancer Using a Radioactive and Fluorescent Tracer; a Feasibility Study
Brief Title: SLN in Colon Cancer Using a Multimodal Tracer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Marjolein Ankersmit, Principal Investigator, VU University of Amsterdam
Allocation: Not Applicable | Model: Single Group
Other Study IDs: NL47648.029.14
Record Dates: First submitted 2016-07-22; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Sentinel Lymph Node
Keywords: colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SLN identification with 89-zirconium-nanocoll (Experimental): Submucosal injection of 2.5 mBq, 0.4 ml 89-Zirconium-Nanocoll and subsequently SLN identification
  Interventions: Procedure: 89Zr-nanocoll and Indocyanine Green

INTERVENTIONS:
Procedure: 89Zr-nanocoll and Indocyanine Green

SUMMARY:
Rationale: Lymph node status is the most important factor in the selection of patients for adjuvant chemotherapy after surgical treatment of primary colorectal carcinoma. Up to 30% stage I/II patients with negative lymph node involvement will develop distant metastases and eventually die from colorectal carcinoma (CRC). Better detection and pathologic staging of the lymph nodes could contribute to a better survival of colon cancer patients. This sentinel lymph node (SLN) procedure aims to identify the first draining lymph node(s) from the primary tumour, which have the highest risk of harbouring metastases. These SLNs can be pathological analysed with several more sensitive histopathologic techniques like immunohistochemical staining (IHC).

Objective: Aim of this study is to investigate if the combination of a radioactive and fluorescent tracer can increase the sensitivity and specificity of the sentinel lymph node mapping (SLNM) technique in colon cancer by utilizing the radioactive component for preoperative imaging (PET/CT) of the SLNs and the near infrared (NIR) fluorescence component for guidance to the SLNs during surgery.

Study design: Single centre pilot study Study population: Ten patients with colon cancer (colon ascendens, colon transversum, colon descendens, sigmoid) stage Tis-T1-T2-T3, scheduled for laparoscopic surgical resection of the tumour.

Intervention (if applicable):

The present study will be performed with the radioactive tracer 89Zr-Nanocoll and fluorescent tracer Indocyanine Green (ICG). A colonoscopy will be performed to inject the radioactive tracer 48 hrs before surgery. After injection, patients will undergo the first PET/CT scan. A second PET/CT scan will be performed ± 24 hrs after tracer injection and a third scan just before the surgical procedure; ± 48 hrs after tracer administration. During the surgical procedure ICG diluted in saline and human albumin will be injected at the base of the tumour by colonoscopy. The PET/CT images will be compared with respect to the total number and location of foci and , if visible, lymphatic vessels. During surgery the fluorescent nodes will be marked with a suture in vivo. Thereafter the PET/CT images will be used as a roadmap, to detect SLNs which are not visible with the NIR laparoscope. These nodes will be marked with a suture too. When all radioactive and/ or fluorescent nodes are detected, the specimen will be resected like the conventional method. Ex vivo the specimen will be inspected for fluorescent and/or radioactive nodes not found in vivo. All the identified nodes will be taken out ex vivo and stored separately. The entire specimen will be submitted for pathologic examination. All identified SLNs will be stained with hematoxylin-eosin (H&E). If the fluorescent or radioactive SLNs are negative after routine H&E staining, they will be sliced in multiple parts and examined with H&E staining and immunohistochemistry with the specific marker CAM5.2. Finally, the pathologist uses palpation to identify the remaining non-fluorescent and/ or radioactive lymph nodes. Nodes found by palpation will be screened for fluorescent and/ or radioactive activity too.

The amount of tumour tissue in positive nodes will be evaluated with the Q-prodit; an interactive video morphometry system (Leica, Cambridge, UK).

Main study parameters/endpoints: Main study parameter is the identification rate of SLN mapping with preoperative PET/CT scans combined with intraoperative near-infrared (NIR) fluorescence imaging in patients with colon carcinoma. Thereby biodistribution and kinetics of 89Zr-Nanocoll have to be considered as primary study parameter. Secondary endpoints are the number and localization of the SLNs and optimal tracer volume.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participating patients will receive conventional resection of the tumour and follow-up according to normal standards in our hospital. The main goal of this study is to optimize the SLN mapping technique in colon cancer. If the investigators are able to identify the true SLN this could lead to better staging and survival of patients with this type of cancer. . Because of the colonoscopy ± 48 hrs before surgery, patients stay in the hospital will be prolonged with one day. The additional risks of exposure to radiation for participating patients are calculated and can be considered as negligible.

ELIGIBILITY:
Inclusion Criteria:

* Oral and written informed consent
* Age 18 years and older
* Colon cancer (Tis-T1-T2-T3)
* Laparoscopic surgical resection of the tumour
* Regular pre-operative work-up

Exclusion Criteria:

* Patients younger than 18 years
* Patients who are legally or mentally incapable or unable to give informed consent
* Gross lymph node involvement
* Invasion of the tumour in surrounding tissue
* Distant metastases
* T4 or metastatic disease discovered during intraoperative staging
* Contraindications to laparoscopic surgery
* Patients at higher risk for anaphylactic reactions
* Pregnancy
* Recent myocardial infarction
* Allergy for iodine
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Identification rate of SLNM with preoperative PET/CT imaging and intraoperative NIR fluorescence imaging in patients with colon carcinoma. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands